CLINICAL TRIAL: NCT03728192
Title: Inhibition and Cytotoxic Effects of Mangosteen on Cell Lines
Brief Title: In-vitro Effect of Mangosteen Pericarp Extract on Cell Lines
Acronym: invitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Director of post graduate studies, Meenakshi Ammal Dental College and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAHER-MU-004-IEC/2016
Record Dates: First submitted 2018-07-13; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Apoptosis
MeSH Terms: interventions — Camptothecin

STUDY DESIGN:
Intervention Model Description: The study comprised of two groups A (Hela) and group B ( H357) . Each group was further subdivided into 3 subgroups- A1 -Untreated cells, A2- mangosteen treated cells and A3- cells treated with standard drug. Group B was divided into B1- Untreated cells, B2- mangosteen treated cells and B3 -cells treated with the standard drug healthy periodontium. Test group: (Chronic periodontitis patients) comprised of 25 participants with signs of clinical inflammation and bone los
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mangosteen treated group (Experimental): HeLa and H357 cell lines were procured and were further subdivided into 2 subdivisions and were assigned interventions:
  Mangosteen group- cells treated with mangosteen extract and Camptothecin group - cells treated with standard anticancer drug camptothecin(25 micro mole)
  Interventions: Other: mangosteen extract
- Untreated group (No Intervention): H357 and HeLa cell line without any drug intervention.

INTERVENTIONS:
Other: mangosteen extract — For Mangosteen group :DNA fragmentation assay is used to identify apoptosis.1×106 cells were harvested and treated with mangosteen pericarp extract for 48 h For Camptothecin group : Cells were also treated with standard anticancer drug Camptothecin to act as a positive control.
  Other Names: camptothecin
  Arms: Mangosteen treated group

SUMMARY:
The present study is an effort to investigate the hypothesis that in-vitro vitality and antiapoptotic effect of alcoholic crude extract of mangosteen on Oral cancer( H357) cell lines and Cevical cancer (HeLa) cell lines.

DETAILED DESCRIPTION:
The oral and cervical cells were investigated by MTT (3-4,5- dimethylthiazol-2-yl)-2,5-diphenyl tetrazolium bromide) assay, DNA fragmentation detection by TUNEL (Terminal deoxynucleotidyl transferase-mediated d-UTP Nick End Labeling) assay and Apototic assay using Annexin V/FITC Kit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral squamous cell carcinoma
* Patients with cervical carcinoma

Exclusion Criteria:

• Patients with leukaemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
apoptotic potential of ethanolic extract of mangosteen pericarp on oral and cervical cancer cell lines via apoptotic assay | 48 hrs at base line
  Apoptosis assay was performed using Annexin V/FITC Kit (BD Biosciences, Catalog no. 556547), and the fluorescence intensities of FITC-conjugated annexin-V and Propidium iodide (PI) in cells were analyzed using flow cytometry. HeLa and H357 cells (1×106 cells/well) were seeded in a 6-well plate. The cells were allowed to adhere for 12 hrs, cultured in medium containing different concentrations of mangosteen extract for 48hr. The cells were then collected and washed twice with Phosphate buffer Saline, gently resuspended in 100μL annexinV-FITC binding buffer (1x) and incubated with 5μL annexinV-FITC in the dark for 10 min at 25°C. This was followed by centrifugation of cells at 2000 rpm for 5 min, and gently resuspended in 500μL annexinV-FITC binding buffer (1x) and 5μL PI was added in an ice bath, followed by immediate analysis by flow cytometry Cell Quest software (BD Biosciences).

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS,PhD, Principal Investigator — Meenakshi academy of higher education and research

IPD SHARING:
Plan to Share IPD: No